CLINICAL TRIAL: NCT00941551
Title: Five-year Follow up of a Randomized Clinical Trial of Unilateral Thyroid Lobectomy With or Without Levothyroxine Treatment Postoperatively
Brief Title: Thyroid Lobectomy With or Without Levothyroxine Treatment Postoperatively
Status: Completed | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Piotr Laider / Head of the Biomedical Research Committee of the Jagiellonian University, Jagiellonian University medical College
Other Study IDs: BBN/501/ZKL/69/L
Record Dates: First submitted 2009-07-16; First posted 2009-07-17 (Estimated); Last update posted 2009-07-17 (Estimated); Status verified 2009-07

CONDITIONS: Recurrent Goiter
Keywords: Thyroid lobectomy,; prophylactic levothyroxine treatment,; recurrent nodular goiter,; iodine deficiency,; long-term follow-up,; completion thyroidectomy
MeSH Terms: conditions — Goiter; Goiter, Nodular | interventions — Thyroxine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group A: receiving levothyroxine postoperatively
  Interventions: Drug: levothyroxine
- Group B: not-receiving levothyroxine postoperatively
  Interventions: Drug: no levothyroxine

INTERVENTIONS:
Drug: levothyroxine — levothyroxine 75-125 ug/day
  Other Names: LT4(+)
  Groups: Group A
Drug: no levothyroxine — observation only without prophylactic levothyroxine
  Other Names: LT4(-)
  Groups: Group B

SUMMARY:
The aim of this study was to compare the prevalence of recurrent nodular goiter in the contralateral thyroid lobe among patients after unilateral thyroid lobectomy for unilateral multinodular goiter receiving versus not receiving prophylactic levothyroxine treatment postoperatively in a five-year follow-up of a randomized study

DETAILED DESCRIPTION:
It is commonly accepted that in patients with benign nodular thyroid disease who undergo operative therapy, surgical resection consists of lobectomy for patients with disease limited to one lobe. Contralateral disease is excluded in such cases by preoperative palpation, ultrasonography of the neck, and intraoperative palpation. On the other hand, the preferred operative procedure for bilateral nodular thyroid disease is total thyroidectomy. Such a treatment strategy minimizes the risk of development of recurrent disease and diminishes the risk of complications when reoperation for recurrent nodular thyroid disease becomes necessary. The recurrence rate for unilateral thyroidectomy of benign nodular goiter performed by expert surgeons has been reported to vary from 10% to 26%. Potential risk factors for recurrence of nodular goiter have been evaluated in many studies and include: young age at presentation, female gender, positive family history of goiter, long duration of symptoms, mutinodularity of thyroid disease, high volume of left thyroid tissue. However, most studies evaluating the incidence of recurrent nodular disease are retrospective, and it is difficult to determine whether the recurrence represents de novo nodule formation in a previously normal thyroid remnant or progression of residual disease left at initial operation.

It is well known fact, that most patients after thyroid lobectomy are euthyroid (60%-90%) and do not require thyroid hormone replacement therapy. However, it is an important question whether thyroid hormone administration postoperatively can prevent recurrent nodular thyroid disease in euthyroid hemithyroidectomized patients? The aim of the present randomized study was to compare the prevalence of recurrent nodular goiter in the contralateral thyroid lobe among patients after unilateral thyroid lobectomy for unilateral multinodular goiter (MNG) receiving versus not receiving prophylactic levothyroxine (LT4) treatment postoperatively in a five-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* unilateral multinodular goiter with normal appearing on ultrasound of the neck contralateral thyroid lobe, in a patient in euthyroid state

Exclusion Criteria:

* bilateral multinodular goiter, enlargement of contralateral thyroid lobe (volume on ultrasound >10 ml), suspicion of thyroid cancer, previous thyroid surgery, thyroiditis, subclinical or clinically overt hypothyroidism or hyperthyroidism, pregnancy or lactation, age < 18 years or > 65 years, ASA 4 grade (American Society of Anesthesiology), and inability to comply with the follow-up protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2000-01; Primary Completion 2003-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Primary outcome measure was prevalence of recurrent goiter within the contralateral thyroid lobe | at 3, 6, 9, 12, 24, 36, 48 and 60 months postoperatively

SECONDARY OUTCOMES:
Secondary outcome was the rate of the reoperation for the recurrent goiter | at 3, 6, 9, 12, 24, 36, 48 and 60 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Marcin Barczynski, MD, PhD, Principal Investigator — Jagiellonian University College of Medicine
Locations (1):
- Jagiellonian University, College of Medicine, Department of Endocrine Surgery, 3rd Chair of General Surgery, Krakow, Poland

REFERENCES:
- [Background] Szybinski Z, Golkowski F, Buziak-Bereza M, Trofimiuk M, Przybylik-Mazurek E, Huszno B, Bandurska-Stankiewicz E, Bar-Andziak E, Dorant B, Kinalska I, Lewinski A, Klencki M, Rybakowa M, Sowinski J, Szewczyk L, Szponar L, Wasik R. Effectiveness of the iodine prophylaxis model adopted in Poland. J Endocrinol Invest. 2008 Apr;31(4):309-13. doi: 10.1007/BF03346363. PMID 18475048
- [Background] Bellantone R, Lombardi CP, Boscherini M, Raffaelli M, Tondolo V, Alesina PF, Corsello SM, Fintini D, Bossola M. Predictive factors for recurrence after thyroid lobectomy for unilateral non-toxic goiter in an endemic area: results of a multivariate analysis. Surgery. 2004 Dec;136(6):1247-51. doi: 10.1016/j.surg.2004.06.054. PMID 15657583
- [Background] Miccoli P, Antonelli A, Iacconi P, Alberti B, Gambuzza C, Baschieri L. Prospective, randomized, double-blind study about effectiveness of levothyroxine suppressive therapy in prevention of recurrence after operation: result at the third year of follow-up. Surgery. 1993 Dec;114(6):1097-101; discussion 1101-2. PMID 8256213
- [Background] Bistrup C, Nielsen JD, Gregersen G, Franch P. Preventive effect of levothyroxine in patients operated for non-toxic goitre: a randomized trial of one hundred patients with nine years follow-up. Clin Endocrinol (Oxf). 1994 Mar;40(3):323-7. doi: 10.1111/j.1365-2265.1994.tb03926.x. PMID 8187295
- [Background] Carella C, Mazziotti G, Rotondi M, Del Buono A, Zito G, Sorvillo F, Manganella G, Santini L, Amato G. Iodized salt improves the effectiveness of L-thyroxine therapy after surgery for nontoxic goitre: a prospective and randomized study. Clin Endocrinol (Oxf). 2002 Oct;57(4):507-13. doi: 10.1046/j.1365-2265.2002.01628.x. PMID 12354133
- [Derived] Barczynski M, Golkowski F, Hubalewska-Dydejczyk A, Konturek A. Twenty-year follow-up of a randomized clinical trial of unilateral thyroid lobectomy with or without postoperative levothyroxine treatment. World J Surg. 2025 Jan;49(1):140-147. doi: 10.1002/wjs.12403. Epub 2024 Nov 15. PMID 39547954